CLINICAL TRIAL: NCT01719731
Title: Psychoeducation of Borderline Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Mary Zanarini, Professor of Psychology, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH095818 (NIH)
Record Dates: First submitted 2012-10-26; First posted 2012-11-01 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Borderline Personality Disorder
Keywords: BPD
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Education (Placebo Comparator): This group will not receive the psychosocial education.
  Interventions: Behavioral: Non-Education
- Education (Active Comparator): This group will receive the psychosocial education
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — This group will receive the psychoeducation
  Arms: Education
Behavioral: Non-Education — This group will not receive the psychoeducation
  Arms: Non-Education

SUMMARY:
Recent research suggests that BPD is a common, serious but treatable disorder with a better than previously recognized prognosis. Despite these findings, many patients with BPD are not given the borderline diagnosis by the mental health professionals treating them. It is also true that many newly diagnosed borderline patients are not provided with up-to-date information on the disorder even though psychoeducation has been found to be a useful form of treatment for other serious psychiatric illnesses.

The investigators have conducted a preliminary randomized trial of psychoeducation for BPD that found that those provided with immediate psychoeducation had a significantly greater reduction in two core symptoms of BPD--general impulsivity and stormy relationships--than those with delayed psychoeducation.

However, both instruction and assessment of change over time were conducted in person by paraprofessionals. The importance of the current study is that it will allow the investigators to develop and test the efficacy of an internet-based program of psychoeducation for BPD that will be both cost efficient and easy to disseminate widely, particularly to underserved populations.

DETAILED DESCRIPTION:
Clinical experience suggests that many people with borderline personality disorder (BPD) are not told of their borderline diagnosis by those treating them. Clinical experience also suggests that many people with newly diagnosed BPD are not provided with up-to-date information on the disorder. These practices are unfortunate as the results of a preliminary, randomized, controlled trial of psychoeducation for BPD conducted by the investigators suggest that informing patients about BPD soon after diagnostic disclosure may be an effective form of early treatment for BPD as it significantly reduced the severity of two of the core symptoms of borderline psychopathology-general impulsivity and unstable relationships.

This application proposes building on the PI's prior work in this area by developing a web-based program for the education of those with BPD and the assessment of three key outcomes; psychoeducation and assessment of outcome that had previously been provided by a team of clinically experienced research assistants. Both of these initiatives would allow for the widespread, cost-efficient dissemination of this early form of treatment for BPD-a form of treatment that has proven effective for other serious psychiatric illnesses.

The investigators first aim is to update our curriculum for teaching individuals with BPD the latest information concerning the disorder. This information will be organized into seven modules: introductory information (history of diagnosis, stigma associated with disorder, and demographic characteristics associated with BPD), symptoms of BPD, co-occurring disorders, etiology, longitudinal course, psychosocial treatments, and psychotropic medications. Some modules will be divided into sub-modules. For example, etiology will encompass childhood adversity, family history of psychiatric disorder, temperament, genetics, and other biological findings.

The investigators second aim is to develop a website for teaching the most up-to-date information about BPD and assessing three key outcomes: the severity of borderline psychopathology, psychosocial impairment, and treatment utilization over time. These outcomes will be assessed using self-report measures with proven psychometric properties. Symptom severity will be accomplished through the internet-based administration of the self-report version of the already widely used Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD)-a dimensional measure of the nine Diagnostic and Statistical Manual of Mental Disorders, fourth edition(DSM-IV) symptoms of BPD. The investigators will also use the Borderline Evaluation of Severity over Time (BEST) developed by Pfohl and Blum as a secondary measure of change in severity of borderline psychopathology. Two other self-report measures will be used to assess psychosocial impairment (Sheehan Disability Scale and Weissman's Social Adjustment Scale). The use of nine forms of psychiatric treatment will be assessed using a self-report version of the treatment section of the Background Information Schedule and its follow-up analog.

The investigators third aim is to conduct a small-scale randomized controlled trial of psychoeducation for BPD using this set of web-based instructional and assessment tools. Half of the 80 subjects will be randomized to the investigators web-based intervention, which will occur a week after diagnostic disclosure, and half will not. The investigators plan to assess symptom severity, psychosocial impairment, and treatment utilization each week for 12 weeks (as the investigators did in our prior study) using the web-based self-report measures described above to determine its immediate effects. The investigators also plan to assess these outcomes using these measures at six months, nine months, and 12 months after randomization to determine if these effects are long lasting. The investigators hypothesize that two of the nine symptoms of DSM-IV BPD will decline significantly more in the subjects who receive psychoeducation than those who do not-general impulsivity and unstable relationships. The investigators further hypothesize that those in the treatment group will have more improved functioning in the social and vocational (but not family realm) than those in the non-treatment group. Finally, the investigators hypothesize that those receiving psychoeducation will be more likely to seek out ongoing psychiatric treatment and less likely to use emergency psychiatric services, such as hospitalizations, than those who do not receive psychoeducation concerning BPD.

If successful, the results of this trial would provide further evidence that psychoeducation is a useful form of early treatment for BPD. These results would also suggest that our web-based platform is an effective and cost efficient method for delivering such a program. Finally, these results would pave the way for a large-scale, multi-site randomized controlled trial of this web-based program in community settings.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18 to 30
* Meets criteria for Borderline Personality Disorder
* Intelligence Quotient must be 71 or higher

Exclusion Criteria:

* Males
* Schizophrenia
* Schizoaffective Disorder
* Bipolar I
* Serious Substance Use Disorder
* Subjects cannot be in treatment at baseline

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Zanarini Rating Scale for Borderline Personality Disorder | Change from baseline through weeks 2-12, 6 month follow-up, 9 month follow-up, 12 month follow-up
  A dimensional self-report measure of the nine DSM-IV symptoms of BPD

SECONDARY OUTCOMES:
Borderline Evaluation of Severity over Time | Change from baseline through weeks 2-12, 6 month follow-up, 9 month follow-up, 12 month follow-up
  A self-report that measures change in severity of borderline psychopathology

OTHER OUTCOMES:
Sheehan Disability Scale | Change from baseline through weeks 2-12, 6 month follow-up, 9 month follow-up, 12 month follow-up
  A self-report measure used to assess psychosocial impairment
Weissman's Social Adjustment Scale | Change from baseline through weeks 4,8,12, 6 month follow-up, 9 month follow-up, 12 month follow-up
  A self-report measure used to assess psychosocial impairment
Clinically Useful Depression Outcome Scale | Change from baseline through weeks 2-12, 6 month follow-up, 9 month follow-up, 12 month follow-up
  A self-report designed to assess sensitivity to change in depression symptoms
Clinically Useful Anxiety Outcome Scale | Change from baseline through weeks 2-12, 6 month follow-up, 9 month follow-up, 12 month follow-up
  A self-report designed to assess sensitivity to change in anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Zanarini, Ed.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Zanarini MC, Conkey LC, Temes CM, Fitzmaurice GM. Randomized Controlled Trial of Web-Based Psychoeducation for Women With Borderline Personality Disorder. J Clin Psychiatry. 2018 May/Jun;79(3):16m11153. doi: 10.4088/JCP.16m11153. PMID 28703950